CLINICAL TRIAL: NCT02991378
Title: Early Intervention Skills for Preschool Children With Emotional and Stress Related Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Shanghai Changning Mental Health Center (Unknown); Putuo Maternal and Child Health Care Hospital (Unknown); Mental Health Center of Shanghai Hongkou District (Unknown); Jingan Maternal and Child Health Care Hospital (Unknown); Maternal and Infant Healthy Center of Hongkou District, Shanghai (Unknown)
Responsible Party: Principal Investigator, Jinsong Zhang, Director of Department of Medical Psychology, Department of Developmental Behavioral and Child Healthcare, Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: XH-16-042
Record Dates: First submitted 2016-11-22; First posted 2016-12-13 (Estimated); Last update posted 2018-04-24 (Actual); Status verified 2018-04

CONDITIONS: Mental Disorder, Child
Keywords: preschool children; emotional disorders/problems; stress related disorders/problems; early intervention
MeSH Terms: conditions — Neurodevelopmental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Subjects in this group will receive the "Children's emotional and stress coping program" which train the children the emotional self-regulation skills and stress coping skill with a standardized protocol.
  Interventions: Behavioral: Children's emotional and stress coping program
- Control group (No Intervention): Subjects in this group will not receive the "Children's emotional and stress coping program".

INTERVENTIONS:
Behavioral: Children's emotional and stress coping program — Giving the children lessons about the emotional self-regulation skills and stress coping skills, with the psychoeducation books and lectures for the teachers and parents.
  Arms: Intervention group

SUMMARY:
This study is about early intervention for preschool children with emotional and stress related disorders. To develop a set of program that could be used in district hospitals for early intervention of preschool children with emotional and stress related disorder or problems.

DETAILED DESCRIPTION:
The objective of this study will be including two aspects. The first one is to develop a set of comprehensive program that including psychoeducation, screening, basic assessment, diagnosis and basic treatment on the emotional and stress related disorders/problems in preschool children. This program is easy implemented for the psychiatrists and pediatricians who work in district primary hospitals. They are not only see patients in hospital but also responsible for the healthcare education in community and kindergarten. In this project they will be trained to master the knowledge and skills on early intervention on the emotional and stress related disorders/problem for preschool children in kindergarten and the basic treatment skills in clinic. The second aspect is the district primary psychiatrists and pediatricians provide psychoeducation, screening and training in kindergarten. The teachers will be trained the program on teaching children the skills on emotional self-regulation and basic stress coping. It's expected that this program will help the primary psychiatrists and pediatricians' clinical skills and help them to improve the awareness and skills of children's emotional and stress related problems/disorder in teachers and parents, improve children's emotional and stress related problems/disorders.

The comprehensive program will include the attained achievements from our past research (the screening questionnaires, interview methods, booklets and protocol for teachers and parents, book and courses for training children on emotional self-regulation and stress coping skills, a simplified CBT manual for children that the trained psychiatrist could use. Xinhua Hospital will be leading this project and 5 primary hospitals in 4 districts will be involved in. These five collaborators hospitals were selected from Shanghai district-level Maternal and Child Health hospitals and district-level Mental Health Center as a pilot.

The selected pediatricians will be major at development and behavioral area, and psychiatrists will be preferring children. They will be trained the common emotional and stress related disorders, screening methods, basic diagnosis skill and basic intervention techniques. After training, they could provide the preventive intervention in kindergarten and the basic service in clinic. Five hundred children from four years old to six years old will be in the early intervention group, and another five hundreds children at the same age will be in the control group for waiting the intervention. The comparisons of the two groups will be on the knowledge improvement in teacher and parents, the decrease of the prevalence of and the level of emotional and stress related disorders/problems.

ELIGIBILITY:
Inclusion Criteria:

* The early intervention for all the children in kindergartens including all the children from four to six years old without severe physical disorders and mental disorders;
* The children who will get the further intervention in hospital should be diagnosed as the childhood emotional disorders and stress related disorders according to ICD-10 diagnostic criteria (International Classification of Diseases 10th) or the children with obvious symptoms but do not fully meet the diagnostic criteria will also be enrolled into the intervention group. The children who have the symptoms after the screening and interview in kindergartens will be refered to hospital.

Exclusion Criteria:

* excluding severe physical disease and neurological developmental disorders can not be participants

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 800 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2018-03-30 (Actual)

PRIMARY OUTCOMES:
level of children's emotional and stress symptoms | through the intervention completion, an average of 2 months
  children's emotional and stress symptoms assessed by children's emotional and stress symptom screening checklist
level of children's positive and negative behaviors | through the intervention completion, an average of 2 months
  children's positive and negative behaviors assessed by Short and long questionnaire for young children
level of chidlren's stress symptoms | through the intervention completion, an average of 2 months
  chidlren's stress symptoms assessed by Stress symptom checklist for children

SECONDARY OUTCOMES:
level of emotional and stress related problems | Six months later after the intervention program completion
  children's emotional and stress symptoms assessed by children's emotional and stress symptom screening checklist
rate of knowledge awareness | through the intervention and psychoeducation completion, an average of 2 months
  the knowledge awareness of teacher and parents on children's emotional and stress problems and management

CONTACTS AND LOCATIONS:
Overall Officials: Jinsong Zhang, PhD, Study Director — Xinhua Hospital, Shanghai Jiao Tong University School of Medicine; Lan Shuai, PhD, Principal Investigator — Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Xinhua Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided